CLINICAL TRIAL: NCT06835127
Title: Feasibility Study of the Use of Ultra-low Dose Iodinated Contrast Agent for Endovascular Procedures in Patients With Chronic Limb-threatening Ischemia and Renal Impairment
Brief Title: Ultra-low Dose Contrast for Endovascular Procedures
Acronym: ULTRA-LOW
Status: Active, not recruiting | Type: Observational
Sponsor: Attikon Hospital (Other)
Responsible Party: Principal Investigator, Stavros Spiliopoulos, Professor of Interventional Radiology, Attikon Hospital
Other Study IDs: ABD126
Record Dates: First submitted 2025-02-12; First posted 2025-02-19 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-11

CONDITIONS: Renal Impairment; Limb Ischemia, Critical
Keywords: Endovascular procedures; Angioplasty; Stenting; Acute kidney injury
MeSH Terms: conditions — Renal Insufficiency; Chronic Limb-Threatening Ischemia; Acute Kidney Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study cohort: Patients with renal disease stages 2-4, scheduled to undergo infrainguinal endovascular procedures due to CLTI, using ultra-low dose of iodine contrast media.
  Interventions: Procedure: Infrainguinal peripheral endovascular revascularization

INTERVENTIONS:
Procedure: Infrainguinal peripheral endovascular revascularization — Percutaneous endovascular angioplasty and/or stenting of infrainguinal arteries (femoropopliteal and/or infrapopliteal arteries) under local anesthesia and adjunct mild conscious sedation.

SUMMARY:
The purpose of this protocol is to study the safety and feasibility of using ultra-low dose iodinated contrast agent for infrainguinal endovascular revascularization procedures in patients with chronic limb-threatening lower limb ischemia (CLTI) and impaired renal function, in the new angiography suite of our department.

DETAILED DESCRIPTION:
Prospective, single-center observational study of patients with CLTI and renal failure but not on dialysis (eGFR <60ml/minute/1.73m2, renal disease stages 2-4), who are scheduled to undergo endovascular revascularization procedures of the lower limb arteries. The procedures will be performed on the new angiograph of the interventional radiology unit (Philips Azurion 7 b20/15 biplane) and the contrast administration protocol will include 1:9 or 2:9 dilutions of iso-osmotic iodinated contrast agent (Visipaque 320mg/ml) with saline, with the aim of administering the minimum possible amount for the safe and effective performance of the procedure (As Low As Possible; ALARA).

ELIGIBILITY:
Inclusion Criteria:

* CLTI
* Prescheduled infrainguinal revascularization procedure
* Renal disease stage 2-4 (eGFR <60ml/minute/1.73m2)
* Adequate pre- and post-procedural hydration protocol

Exclusion Criteria:

* Inadequate pre- and post-procedural hydration protocol
* End-stage renal disease/ dialysis
* eGFR >60ml/minute/1.73m2)
* Endovascular treatment of Iliac artery steno-oclussive disease
* Allergy to contrast media

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients suffering from renal impairment stage 2 to 4 and chronic -limb-threatening ischemia (CLTI)
Sampling Method: Non-Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2024-09-01 (Actual); Primary Completion 2026-01-23 (Estimated); Study Completion 2026-01-23 (Estimated)

PRIMARY OUTCOMES:
Renal function | From the end of the procedure to day 2
  Assessment of eGFR
Technical success | Day 1
  Successful, uneventful revascularization using less than 15 ml of iodinated contrast media.

SECONDARY OUTCOMES:
Renal function | 1 month
  Introduction in dialysis
Limb salvage | 6 months
  Non pre-scheduled above the knee amputation
Survival | 6 months
  Patients' survival rate
Re-intervention | 6 months
  Target lesion reintervention (TLR) due to clinical deterioration or relapse of symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Stavros C Spiliopoulos, MD, PhD, Principal Investigator — ATTIKO University Hospital
Locations (1):
- "ATTIKON" University General Hospital, , 1st Rimini St,, Chaïdári, Attica, Greece

IPD SHARING:
Plan to Share IPD: Undecided
All study data will be available upon reasonable request

REFERENCES:
- [Background] Conte MS, Bradbury AW, Kolh P, White JV, Dick F, Fitridge R, Mills JL, Ricco JB, Suresh KR, Murad MH, Aboyans V, Aksoy M, Alexandrescu VA, Armstrong D, Azuma N, Belch J, Bergoeing M, Bjorck M, Chakfe N, Cheng S, Dawson J, Debus ES, Dueck A, Duval S, Eckstein HH, Ferraresi R, Gambhir R, Gargiulo M, Geraghty P, Goode S, Gray B, Guo W, Gupta PC, Hinchliffe R, Jetty P, Komori K, Lavery L, Liang W, Lookstein R, Menard M, Misra S, Miyata T, Moneta G, Munoa Prado JA, Munoz A, Paolini JE, Patel M, Pomposelli F, Powell R, Robless P, Rogers L, Schanzer A, Schneider P, Taylor S, De Ceniga MV, Veller M, Vermassen F, Wang J, Wang S; GVG Writing Group for the Joint Guidelines of the Society for Vascular Surgery (SVS), European Society for Vascular Surgery (ESVS), and World Federation of Vascular Societies (WFVS). Global Vascular Guidelines on the Management of Chronic Limb-Threatening Ischemia. Eur J Vasc Endovasc Surg. 2019 Jul;58(1S):S1-S109.e33. doi: 10.1016/j.ejvs.2019.05.006. Epub 2019 Jun 8. PMID 31182334
- [Background] van der Molen AJ, Reimer P, Dekkers IA, Bongartz G, Bellin MF, Bertolotto M, Clement O, Heinz-Peer G, Stacul F, Webb JAW, Thomsen HS. Post-contrast acute kidney injury - Part 1: Definition, clinical features, incidence, role of contrast medium and risk factors : Recommendations for updated ESUR Contrast Medium Safety Committee guidelines. Eur Radiol. 2018 Jul;28(7):2845-2855. doi: 10.1007/s00330-017-5246-5. Epub 2018 Feb 9. PMID 29426991
- [Background] Jens S, Schreuder SM, De Boo DW, van Dijk LC, van Overhagen H, Bipat S, Koelemay MJ, Reekers JA. Lowering iodinated contrast concentration in infrainguinal endovascular interventions: a three-armed randomized controlled non-inferiority trial. Eur Radiol. 2016 Aug;26(8):2446-54. doi: 10.1007/s00330-015-4109-1. Epub 2015 Dec 2. PMID 26630997